CLINICAL TRIAL: NCT00038636
Title: A Study of Two Different Doses of ABT-378/Ritonavir in HIV-Infected Patients Who Have Taken Protease Inhibitors and Non-Nucleoside Reverse Transcriptase Inhibitors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M99-049; NCT00006210 (obsolete NCT alias)
Record Dates: First submitted 2002-06-03; First posted 2002-06-04 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2006-08

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; Ritonavir

INTERVENTIONS:
Drug: Lopinavir/ritonavir
Drug: Ritonavir

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of a high dose of ABT-378/ritonavir

ELIGIBILITY:
Inclusion:

* HIV positive
* Are at least 18 years old
* Subject has not been treated for an active AIDS-defining opportunistic infection within 15 days of screening
* HIV RNA level > 1000 copies/mL
* Previous therapy with at least one protease inhibitor, at least one non-nucleoside reverse transcriptase inhibitor and at least one nucleoside reverse transcriptase inhibitor

Exclusion:

* Subject is pregnant or breast-feeding
* Subject has received an investigational drug within 30 days prior to screening
* Have a history of pancreatitis
* History of intolerance to ritonavir
* Abnormal laboratory tests at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2000-09

PRIMARY OUTCOMES:
Virologic and immunologic activity evaluations include plasma HIV RNA, CD4 and CD8 cell counts

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Sun, M.D., Study Chair — Divisional Vice President, Infectious Diseases and Virology Dept.
Locations (7):
- United States (3):
  - UCSD Treatment Center, San Diego, California
  - Johns Hopkins Hospital, Baltimore, Maryland
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
- France (2):
  - Hopital Pitie-Salpetriere, Paris
  - Hospital Europeen Georges Pompidou, Paris
- Spain (2):
  - Hospital Clinico de Barcelona, Barcelona
  - Ciutat Sanitaria de Bellvitge, Barcelona